CLINICAL TRIAL: NCT02182089
Title: Measuring Cardiovascular Stress in Patients on Hemodialysis Study II
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Intelomed, Inc. (Industry)
Collaborators: Tufts Medical Center (Other); Dialysis Clinic, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: IntelomedTufts11231
Record Dates: First submitted 2014-05-09; First posted 2014-07-08 (Estimated); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: Hypotension of Hemodialysis; Hypotension; Estimated Dry Weight; Myocardial Injury; Arrhythmia
MeSH Terms: conditions — Hypotension; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Dialysis patients with greater than 20% IDH: Study Population:
  The sample will be enriched for subjects prone to IDH, defined as patients who experience IDH for greater than 20% of HD treatments in the past 2 months. The study population will consist of 48 patients total, 75% of patients (n=36) prone to IDH and 25% of patients with less than 10% of IDH during the last two months (n=12).
- Patients with less than 10% IDH: Study Population:
  The sample will be enriched for subjects prone to IDH, defined as patients who experience IDH for greater than 20% of HD treatments in the past 2 months. The study population will consist of 48 patients total, 75% of patients (n=36) prone to IDH and 25% of patients with less than 10% of IDH during the last two months (n=12).

SUMMARY:
The overall goal is to evaluate the predictive accuracy of a measure of autoregulatory adequacy derived from CVInsight and compare it with other measures in recognizing hypotensive events during hemodialysis..

DETAILED DESCRIPTION:
Specific Aims are as follows:

1. Assess the accuracy of a new rule set for CVInsight® in predicting intradialytic hypotensive episodes.
2. Assess the comparative predictive accuracy of CVInsight® to other measures with regard to intradialytic hypotensive events.
3. Assess estimated dry weight goals by monitoring post-dialytic vascular refill using CVInsight® and other measures.
4. Assess hemodialysis(HD)-induced myocardial injury by monitoring the occurrence and frequency of arrhythmias and the levels of cardiac Troponin T.

ELIGIBILITY:
Inclusion Criteria:

Eligibility shall consist of the following:

* Age ≥ 20 years old
* Speaks and understands English, Spanish or Chinese
* Provides Informed Consent
* Patients with 20% intradialytic hypotensive events over the last two months.

Exclusion criteria for both groups:

* Unstable hemodialysis patients per judgment of the clinician prior to the start of the treatment
* Patients unable to have blood pressure cuff measured on the upper arm
* Inability to wear monitor on forehead
* Patients treated with sodium or ultrafiltration profiling and the patient's nephrologist is unwilling to alter this for the study treatments
* Patients unwilling to shave the anterior chest
* Patients with active infection of the upper chest wall tissue.
* Patients with a deep brain stimulator, as it may disrupt the quality of the ECG data.
* Patients who are unwilling to take short showers versus bathing during the 7 day period .
* Patients who require intradialytic testing (ie transonic) during the monitored treatment.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study Population:
  The sample will be enriched for subjects prone to IDH, defined as patients who experience IDH for greater than 20% of HD treatments in the past 2 months. The study population will consist of 48 patients total, 75% of patients (n=36) prone to IDH and 25% of patients with less than 10% of IDH during the last two months (n=12).
Sampling Method: Non-Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2014-04; Primary Completion 2023-03-01 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
Number of intradialytic hypotensive (IDH) episodes that can be detected by the new rule set for CVInsight. | 3-4 hours, for two hemodialysis session, or 6-8 hours total
  IDH defined by at least one of the following: 1) Symptoms of hypotension: dizziness, cramping, altered consciousness, nausea +/- vomiting (new since beginning of session), chest pain, shortness of breath, seizure, diaphoretic. 2) Intervention administered due to IDH; relevant interventions:a) a reduction in ultrafiltration (UF) goal programmed at start of treatment (tx); b) admin. of IV fluid, e.g. saline, mannitol or hypertonic saline; c) stopping tx early due to IDH symptoms or event. 3) A significant drop in blood pressure, regardless of symptoms, defined as:
  * For pts w/ a pre-dialysis systolic blood pressure (SBP) >110 mm Hg, an intra or post-dialysis SBP <90 mm Hg, or a drop of >40 mm Hg over 30 min.
  * For pts w/ a pre-dialysis SBP <110, a decline in SBP <85 mm Hg or 15 mm Hg or lower than their starting BP.

SECONDARY OUTCOMES:
The comparative, predictive accuracy of CVInsight® and CRIT-LINE III with regard to intradialytic hypotensive events. | 3-4 hours, for two hemodialysis session, or 6-8 hours total
  CVInsight® and CRIT-LINE III will have different predictive accuracies in recognizing IDH episodes.
  Receiver Operator Characteristics analysis of CVInsight and CRIT-LINE
  CVInsight: Event level thresholds will be triggered based upon new proprietary rule set.
  CRIT-LINE: Change in hematocrit of 8% per hour or 15% over the treatment.
Amount of post-dialytic vascular refill as separately indicated by both CVInsight® and CRIT-LINE III. | At the end of each dialysis session after the ultrafiltration rate (UFR) has turned off.
  Post-dialytic vascular refill will indirectly reflect hydration status and accuracy of dry weight estimation. Vascular refill -Ten minutes prior to the end of treatment, with UFR at zero, and BFR at same rate as during treatment, measurements will continue to be taken via the CVInsight® and CRIT-LINE devices to assess vascular refill.
  CVInsight: Increase in pulse amplitude.
  CRIT-LINE: Increase of 0.5% increase in hematocrit (HCT) over 10 minutes.
The occurrence and frequency of arrhythmias as indicated on the Zio ECG Patch and the levels of cardiac Troponin T, taken prior to each HD treatment. which are indicative HD-induced myocardial injury.. | 24 hours before first session of monitored dialysis to at least 24 hours after the second session on monitored dialysis sessions.
  Arrhythmias frequency overall, on dialysis days, during long and short interdialytic periods, nocturnal, diurnal. Troponin T levels will correlate with the incidence rates of arrhythmias. Troponin T as measured by ng/mL, reference value at <0.011

CONTACTS AND LOCATIONS:
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States